CLINICAL TRIAL: NCT02880098
Title: Variations of High Sensitivity Troponin T in Neonates
Acronym: TnTc-us
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1615
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Newborn; Newborn, Transient
Keywords: Neonatology; Troponin T; Standards

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Troponin T blood level — assess Troponin T blood level for every child born from the same sample of blood (after clamping the umbilical cord) used for assessment of pH and lactate.

SUMMARY:
Troponin T-us is a cardiac marker for myocardial infarction. Its use in neonates is increasing, yet normal values are still to be determined for the latest generation of tests, such as High sensitivity cardiac troponin T test. This study is an observational study designed to determine biological normal values of High sensitivity cardiac troponin T test (troponin T -us) in newborns.

DETAILED DESCRIPTION:
* Approximately 400 subjects will be recruited over a planned recruitment period of 2 months. During labour, or pre natal hospitalization, information about the study will be given to every mothers by the midwife or the pediatrician. Absence of opposition will be notified in the medical file.
* At birth, every child born alive is possibly eligible for this study, if he doesn't meet the exclusion criteria.
* After clamping the umbilical cord, the midwife realizes the systematic sample for assessment of pH and lactate. If the mother did not object to the study, the midwife will use 200µl of this very same sample to assess Troponin T blood level. This sample goes to the same laboratory to be analyzed. The blood sample for troponin T measurement must be brought to the laboratory within 2 hours, just as pH and lactate must be. The midwife in charge of this patient also fills a form with informations from the patient's medical file. This form is anonymized for the study.
* Samples will not be stored, remaining swab after analysis will be destructed.
* Before discharge, all children undergo a medical exam by a pediatrician, whether they are in maternity or in neonate. The pediatrician who examines the child fills a second form that summarizes the noteworthy events of his hospital journey.

Subjects have the right to withdraw from the study at any time for any reason. If one of the parents wishes to withdraw from the study after the first Troponin T measurement is made, we will ask for their permission to use the collected data.

ELIGIBILITY:
Inclusion Criteria:

* Every newborn, born alive in René Dubos maternity, without regarding the way of birth.
* Absence of malformative syndromes or genetic abnormalities in prenatal echographies
* Absence of parental opposition

Exclusion Criteria:

* Multiple pregnancies
* Post natal discovery of malformative syndromes or genetic abnormality. All congenital heart diseases will be excluded.
* Parental opposition at any time of the study

Ages: 1 Day to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born in hospital René Dubos
Sampling Method: Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2016-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Level of cardiac high sensitive Troponin T in umbilical cord blood | At birth - Time 0
  T level will be analyzed by the biochemistry laboratory and collected by a study investigator.

SECONDARY OUTCOMES:
Noticeable events during pregnancy ; Delivery conditions | Within the two hours following birth
  Any event, disease, treatment during pregnancy. Those data will be collected in the mothers pregnancy file.
Noticeable events in post partum | Before discharge
  Infection, jaundice… Those data will be collected in the baby's maternity file or intensive care unit file

CONTACTS AND LOCATIONS:
Overall Officials: BORRHOMEE Suzanne, PH, Principal Investigator — suzanne.borrhomee@gmail.com
Locations (1):
- CH Rene Dubos, Pontoise, Val d'Oise, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lefevre G. [Troponins: biological and clinical aspects]. Ann Biol Clin (Paris). 2000 Jan-Feb;58(1):39-48. French. PMID 10673613
- [Background] Adamcova M. Troponins in children and neonates. Acta Paediatr. 2003 Dec;92(12):1373-5. doi: 10.1080/08035250310007637. PMID 14971783
- [Background] Fortunato G, Carandente Giarrusso P, Martinelli P, Sglavo G, Vassallo M, Tomeo L, Rea M, Paladini D. Cardiac troponin T and amino-terminal pro-natriuretic peptide concentrations in fetuses in the second trimester and in healthy neonates. Clin Chem Lab Med. 2006;44(7):834-6. doi: 10.1515/CCLM.2006.144. PMID 16776629
- [Background] Nomura RM, Ortigosa C, Fiorelli LR, Liao AW, Zugaib M. Gender-specific differences in fetal cardiac troponin T in pregnancies complicated by placental insufficiency. Gend Med. 2011 Jun;8(3):202-8. doi: 10.1016/j.genm.2011.05.001. PMID 21664586